# **Official Title of the Study**

Strategic Daytime Napping Enhances Agility and Lowers Perceived Exertion but Does Not Improve Fatigue Resistance in Adolescent Soccer Players

ClinicalTrials.gov Identifier NCT: Not yet assigned

Document Type
Study Protocol and Ethics Approval (in Turkish)

This document corresponds to the ClinicalTrials.gov registration record for this study

Document Date 10 May 2025

# Strategic Daytime Napping Enhances Agility and Lowers Perceived Exertion but Does Not Improve Fatigue Resistance in Adolescent Soccer Players

#### DETAILED TRIAL PROTOCOL

#### 1. Structured Abstract

**Background and rationale:** Strategic daytime napping (25 min, 45 min) may acutely influence anaerobic performance in team sports via sleepiness-recovery dynamics.

**Objectives and hypotheses:** Primary objective is to test whether nap conditions improve proagility performance. Hypothesis: N25 and/or N45 outperform N0 on pro-agility time. Secondary objectives examine effects on RSA, RPE, Hooper wellness, and VAS alertness/sleep quality. Exploratory objective assesses associations of PSQI and POMS with outcomes.

**Design:** Quasi-experimental, repeated-measures crossover with 3 conditions (N0, N25, N45), 48-h washout, afternoon sessions, testing 60 min post-awakening.

**Participants and setting:** Sixteen competitive male soccer players (U17–U19), isolated dark rooms at ≈22°C; standardized field/lab conditions.

**Interventions:** N0, 25-min, 45-min nap opportunities; sleep—wake verification by Visual Analogue Scale; prohibition of visual/stimulating activities; standardized warm-up monitored by Polar H10.

**Primary/secondary outcomes:** Primary: Pro Agility Test time. Secondary: RSA (6×30 m, 20-s recovery), RPE, Hooper Index, VAS. Exploratory: correlations with PSQI/POMS.

**Sample size:** G\*Power 3.1.9.7 for RM-ANOVA ( $\alpha$ =0.05, 1- $\beta$ =0.80, f=0.30-0.40) indicated  $\geq$ 12; n=16 recruited.

**Randomization and blinding:** Within-subject random order of conditions; automated timing to reduce measurement bias; assessor blinding not implemented.

Statistical analysis (summary): RM-ANOVA with Bonferroni adjustments; assumption checks (Levene, Mauchly, Greenhouse–Geisser); effect sizes (ηp², Cohen's dz, 95% CI); Pearson correlations.

#### 2. Objectives and Testable Hypotheses

**Primary objective:** Determine whether agility, perceived exertion and fatigue resistence differs between N0, N25, and N45 conditions.

**Primary hypothesis:** N25 and/or N45 conditions gives better results than N0.

**Secondary objectives:** Assess condition effects on Pro Agility time, RSA metrics (best/mean time, fatigue index), RPE, Hooper Index, and VAS alertness/sleep quality.

**Exploratory objectives:** Examine associations between PSQI/POMS and performance/subjective outcomes.

## 3. Study Design

- **Design:** Quasi-experimental, repeated-measures crossover.
- Conditions: N0 (no nap), N25 (25 min), N45 (45 min).
- Order: Randomized within participant.
- Washout: 48 h between sessions [1].
- **Timing:** Nap starts at 14:00; testing begins 60 min post-awakening [2,3].
- **Testing flow:** Warm-up  $\rightarrow$  Pro Agility  $\rightarrow$  3-min rest  $\rightarrow$  RSA; RPE after each sprint.

## 4. Setting and Infrastructure

- Sleep environment: Isolated, ventilated, dark rooms with blackout curtains; ambient temperature ≈22°C [4].
- **Sleep monitoring:** Visual Analogue Scale for sleep—wake verification [5,6].
- **Physiological monitoring:** Polar H10 for heart rate during warm-up [7].

## 5. Participants

#### 5.1 Inclusion Criteria

- Competitive male players from Yeni Malatyaspor U17 or U19 squads.
- Healthy, no recent illness or injury.
- No habitual daytime napping.

#### 5.2 Exclusion Criteria

- Active infection.
- Diagnosed hyperactivity or sleep disorder.
- Experiencing sleep problems on protocol days.
- Non-adherence to instructions, inability to complete sessions, or cooperation issues.

## 5.3 Sampling and Screening

- End-of-season volunteer recruitment from U17–U19 squads.
- Pre-screening by trained staff; verification with training logs.

## **5.4 Informed Consent**

- Written consent from all participants; for those under 18, parental/legal guardian consent obtained.
- Ethics approval: Inonu University Non-Interventional Clinical Research Ethics Committee (Approval No: 2024/5635; Date: 05/03/2024); study conducted in accordance with the Declaration of Helsinki.

#### 6. Interventions

- **Conditions:** N0, N25, N45.
- Nap procedure: 10-min room adaptation at 13:50 [8]; nap opportunity at 14:00; preferred lying position allowed.
- **Verification:** Sleep onset, duration, and awakening verified via Visual Analogue Scale; wakefulness confirmed in N0 [5,6].
- **Pre-session standards:** Avoid strenuous training for 24 h; avoid alcohol for 24 h and caffeine for 6 h; verbal compliance check at arrival [9–11].
- **Prohibited activities:** No phone use, video games, or visually stimulating tasks during all conditions [12,13].
- **Warm-up standardization:** Light jogging plus a 3-min mobility sequence; heart rate monitored with Polar H10 [7].
- **Testing order:** Pro Agility  $\rightarrow$  3-min rest  $\rightarrow$  RSA; RPE recorded after each sprint.

#### 7. Outcomes and Assessment Schedule

## 7.1 Primary Outcome

• Pro Agility Test time (20-yard shuttle, total 18.28 m): Privided agility outcomes [14].

#### 7.2 Secondary Outcomes

- RSA (6×30 m, 20-s recovery): Best/mean time and fatigue index [15–17].
- RPE (Borg 6–20): Recorded after each sprint; session mean used for analysis [18].
- **Hooper Index:** Fatigue, stress, muscle soreness (1–7), sleep quality (1–7) [19].
- VAS (sleep quality and alertness): 0–10 cm and 0–100 mm scales [8].

#### 7.3 Exploratory Outcomes

• **Correlations** of PSQI and POMS with performance and subjective measures (Pearson r) [20–23].

#### 7.4 Schedule of Assessments (Timeline)

| Time point | Screening | T0<br>(Baseline) | Intervention | T1 (60 min post-<br>awakening) |
|---|---|---|---|---|
| Eligibility and consent | X | | | |
| MEQ/PSQI/POMS | | X | | |
| Nap (N0/N25/N45) | | | X | |
| Pro Agility | | | | X |
| RSA + RPE | | | | X |

| Time point | Screening | T0<br>(Baseline) | Intervention | T1 (60 min post-<br>awakening) |
|---|---|---|---|---|
| Hooper | | | | X |
| VAS | | | | X |

#### 8. Sample Size and Justification

- **Software and model:** G\*Power 3.1.9.7; repeated-measures ANOVA (within-subjects, 3 conditions) [24].
- **Parameters:**  $\alpha$ =0.05, 1- $\beta$ =0.80; expected effect size f=0.30-0.40 based on prior literature [9,25,26].
- **Result:** Minimum ≥12; **n=16** recruited to accommodate variability and potential attrition.
- **Note:** Crossover design increases power by using each participant as own control [10].

## 9. Randomization, Allocation Concealment, and Blinding

- Randomization: Within-subject random assignment of condition order.
- **Allocation concealment:** Condition order not disclosed to participants until session day; administered by study staff.
- **Blinding:** Participant blinding is infeasible; automated timing reduces measurement bias; assessor blinding not implemented.
- Unblinding: Not applicable.

#### 10. Study Workflow and Procedures

- 1. **Screening and baseline:** Eligibility, informed consent, demographics and anthropometry (SECA stadiometer; Toledo 2096 PP scale; BMI=kg/m² [27]). MEQ, PSQI, POMS administered once at baseline [20–22,28].
- 2. **Pre-session standards:** 24 h no heavy training; 24 h no alcohol; 6 h no caffeine; verbal verification at arrival [9,11,29].
- 3. **Nap session:** 13:50 adaptation; 14:00 N0/N25/N45; dark quiet room ≈22°C; subjective verification [5,6]; prohibition of visual/stimulating activities [12,13].
- 4. **Warm-up:** Light jog plus 3-min mobility; heart rate monitored with Polar H10 for standardization [7].
- 5. **Performance tests:** 60 min post-awakening [2,3], Pro Agility  $\rightarrow$  3-min rest  $\rightarrow$  RSA (6×30 m, 20-s intervals [15–17]); RPE after each sprint [18].
- 6. **Post-session:** Hooper and VAS forms [8,19].

## 11. Data Collection Instruments and Quality Assurance

- **Devices:** SECA® stadiometer; Toledo 2096 PP scale; 16x Polar H10.
- Validity/reliability: MEQ, PSQI, POMS are validated instruments [20–22,28]; SmarTracks offers high temporal resolution; literature supports actigraphy-based sleep—wake verification with Fitbit [5,6].
- **Staff training:** Test administrators trained before data collection; measurement repeatability monitored.

#### 12. Data Management

- Coding and de-identification: Participant IDs (e.g., P001–P016); personal data stored separately and encrypted.
- Entry and verification: Electronic CRFs; double checks and random source data verification.
- **Missing data:** Multiple imputation may be applied when appropriate; sensitivity analyses reported.
- Access and retention: Restricted to authorized researchers; retention per regulations.

#### 13. Statistical Analysis Plan

- **Software:** SPSS v29.
- **Descriptives:** Mean±SD, min-max.
- Assumption checks: Normality (skewness/kurtosis within  $\pm 1.5$ ), homogeneity (Levene), sphericity (Mauchly; Greenhouse–Geisser corrections if violated).
- **Primary analysis:** RM-ANOVA across N0–N25–N45; Bonferroni where appropriate.
- Effect sizes:  $\eta p^2$  (small <0.06; medium 0.06–<0.14; large  $\ge$ 0.14) and Cohen's dz for pairwise comparisons; 95% CIs [10,30].
- **Secondary analyses:** RM-ANOVA for RSA metrics, RPE, Hooper, and VAS with appropriate corrections.
- **Exploratory analyses:** Pearson correlations between PSQI/POMS and outcome variables [23].
- Missing data and sensitivity: Pre-specified sensitivity checks reported.
- **Pre-specified subgroups:** None; all participants classified as intermediate chronotype (MEQ) [20,28].

#### 14. Safety Monitoring and Adverse Event Management

- **Risk profile:** Low-risk procedures involving brief naps and field-based anaerobic tests.
- **Adverse events:** Monitor for syncope, dizziness, musculoskeletal issues; medical evaluation as needed.

• **Reporting:** Serious adverse events reported within 24 h to the ethics committee per institutional policies.

#### 15. Ethical Considerations

- Ethics approval: Inonu University Non-Interventional Clinical Research Ethics Committee; Approval No: 2024/5635; Date: 05/03/2024.
- Participant rights: Voluntary participation, right to withdraw at any time, confidentiality and data protection per applicable law.
- Conflicts of interest and funding: The authors declare no conflicts of interest.

## 16. Dissemination and Data Sharing Policy

- **Reporting:** Results will be reported in a peer-reviewed journal with a CONSORT flow diagram will be provided in the final report.
- **Data/code sharing:** De-identified data and analysis code to be shared per journal policies and institutional regulations.

#### 17. Timeline and Gantt Plan

- **Preparation (Months 0–1):** Ethics approval, device calibration, staff training, pilot tests.
- Data collection (Months 2–3): Three sessions per participant, 48-h washout.
- Analysis (Months 3–4): Data cleaning, statistical analyses, sensitivity checks.
- Reporting (Months 4–5): Manuscript and supplementary materials.

#### 18. Budget and Resources (optional)

- **Equipment:** SECA stadiometer, Toledo scale, Polar H10.
- Consumables and personnel: Forms, printing, staff time.

#### 19. References

- 1. Ammar, A. *et al.* The effect of a daytime 60-min nap opportunity on postural control in highly active individuals. *Biol Sport* 38, 683–691 (2021).
- 2. Ammar, A. *et al.* Effects of pomegranate supplementation on exercise performance and post-exercise recovery in healthy adults: a systematic review. *British Journal of Nutrition* 120, 1201–1216 (2018).
- 3. Botonis, P. G., Koutouvakis, N. & Toubekis, A. G. The impact of daytime napping on athletic performance A narrative review. *Scand J Med Sci Sports* 31, 2164–2177 (2021).
- 4. Romyn, G. *et al.* Daytime naps can be used to supplement night-time sleep in athletes. *Chronobiol Int* 35, 865–868 (2018).
- 5. Migueles, J. H. *et al.* Accelerometer Data Collection and Processing Criteria to Assess Physical Activity and Other Outcomes: A Systematic Review and Practical Considerations. *Sports Medicine* 47, 1821–1845 (2017).
- 6. Lee, J.-M., Byun, W., Keill, A., Dinkel, D. & Seo, Y. Comparison of Wearable Trackers' Ability to Estimate Sleep. *Int J Environ Res Public Health* 15, 1265 (2018).

- 7. Li, M. & Kim, Y. Design of a Wireless Sensor System with the Algorithms of Heart Rate and Agility Index for Athlete Evaluation. *Sensors* 17, 2373 (2017).
- 8. Souabni, M. *et al.* Napping and heart rate variability in elite athletes. *Biol Sport* 41, 213–221 (2024).
- 9. Romdhani, M. *et al.* The effect of post-lunch napping on mood, reaction time, and antioxidant defense during repeated sprint exercice. *Biol Sport* 38, 629–638 (2021).
- 10. Cohen, J. Statistical Power Analysis for the Behavioral Sciences. (Routledge, 1988).
- 11. Reichert, C. F., Deboer, T. & Landolt, H. Adenosine, caffeine, and sleep-wake regulation: state of the science and perspectives. *J Sleep Res* 31, (2022).
- 12. Kaida, K., Takahashi, M. & Otsuka, Y. A Short Nap and Natural Bright Light Exposure Improve Positive Mood Status. *Ind Health* 45, 301–308 (2007).
- 13. Stowe, S. R., LeBourgeois, M. K. & Diniz Behn, C. Modeling the Effects of Napping and Non-napping Patterns of Light Exposure on the Human Circadian Oscillator. *J Biol Rhythms* 38, 492–509 (2023).
- 14. Göral, K., Hadi, G. & Kaplan, T. Investigation of Futsal Players' Answers to Different Agility Tests According to Their Positions. *Spor ve Performans Araştırmaları Dergisi* 14, 115–126 (2023).
- 15. Wragg, C. B., Maxwell, N. S. & Doust, J. H. Evaluation of the reliability and validity of a soccer-specific field test of repeated sprint ability. *Eur J Appl Physiol* 83, 77–83 (2000).
- 16. Dawson, B. Repeated-Sprint Ability: Where Are We? *Int J Sports Physiol Perform* 7, 285–289 (2012).
- 17. Schimpchen, J., Skorski, S., Nopp, S. & Meyer, T. Are "classical" tests of repeated-sprint ability in football externally valid? A new approach to determine in-game sprinting behaviour in elite football players. *J Sports Sci* 34, 519–526 (2016).
- 18. Vitale, J. A. & Weydahl, A. Chronotype, Physical Activity, and Sport Performance: A Systematic Review. *Sports Medicine* 47, 1859–1868 (2017).
- 19. Hsouna, H. *et al.* Effect of different nap opportunity durations on short-term maximal performance, attention, feelings, muscle soreness, fatigue, stress and sleep. *Physiol Behav* 211, 112673 (2019).
- 20. Núñez, P., Perillan, C., Arguelles, J. & Diaz, E. Comparison of sleep and chronotype between senior and undergraduate university students. *Chronobiol Int* 36, 1626–1637 (2019).
- 21. Selvi, Y., Gulec, M., Aydin, A. & Besiroglu, L. Psychometric evaluation of the Turkish language version of the Profile of Mood States (POMS). *Journal of Mood Disorders* 1, 152 (2011).
- 22. Petrowski, K., Albani, C., Zenger, M., Brähler, E. & Schmalbach, B. Revised Short Screening Version of the Profile of Mood States (POMS) From the German General Population. *Front Psychol* 12, (2021).
- 23. Bakdash, J. Z. & Marusich, L. R. Repeated Measures Correlation. *Front Psychol* 8, (2017).

- 24. Faul, F., Erdfelder, E., Lang, A.-G. & Buchner, A. G\*Power 3: A flexible statistical power analysis program for the social, behavioral, and biomedical sciences. *Behav Res Methods* 39, 175–191 (2007).
- 25. Romdhani, M. *et al.* Improved Physical Performance and Decreased Muscular and Oxidative Damage With Postlunch Napping After Partial Sleep Deprivation in Athletes. *Int J Sports Physiol Perform* 15, 874–883 (2020).
- 26. Souabni, M., Hammouda, O., Souabni, M. J., Romdhani, M. & Driss, T. 40-min nap opportunity attenuates heart rate and perceived exertion and improves physical specific abilities in elite basketball players. *Research in Sports Medicine* 31, 859–872 (2023).
- 27. Sales, M. *et al.* Vertical Jump Is Strongly Associated to Running-Based Anaerobic Sprint Test in Teenage Futsal Male Athletes. *Sports* 6, 129 (2018).
- 28. Özdalyan, F., Tütüncü, Ö., Gümüş, H. & Açıkgöz, O. Reliability and Validity of the Turkish Version of the Morningness Eveningness Questionnaire. *Neurological Sciences and Neurophysiology* 38, 50–59 (2021).
- 29. Hudson, A. N., Van Dongen, H. P. A. & Honn, K. A. Sleep deprivation, vigilant attention, and brain function: a review. *Neuropsychopharmacology* 45, 21–30 (2020).
- 30. Richardson, J. T. E. Eta squared and partial eta squared as measures of effect size in educational research. *Educ Res Rev* 6, 135–147 (2011).

## T.C. İNÖNÜ ÜNİVERSİTESİ BİLİMSEL ARAŞTIRMA VE YAYIN ETİĞİ KURULU (Sağlık Bilimleri Girişimsel Olmayan Klinik Araştırmalar Etik Kurulu)

| Oturum Tarihi | Oturum Sayısı | Karar Sayısı |
|---|---|---|
| 05.03.2024 | 05 | 2024/5635 |
| Çalışma Adı | Futbolcularda Stratejik Şekerlemenin Bazı Anaerobik Performanslara<br>Etkisi: Kronotip Açısından Değerlendirme | |
| Araştırmacılar | Doç. Dr. Özgür EKEN ( Yürütücü )<br>Yükseklisans Öğrencisi Mertkan ÖNCÜ ( Yardımcı Araştırmacı ) | |

Başvurunuz; üniversitemiz Bilimsel Araştırma ve Yayın Etiği Yönergesi açısından uygun olupolmadığı hususundaki başvurusuna ilişkin raportör raporu görüşüldü. Çalışma Bilimsel Araştırma ve Yayın Etiği Yönergesi açısından değerlendirildiğinde *çalışmanın etik açıdan uygun olduğuna*; oy birliği ile karar verilmiştir.

> ASLI CARANA Gamzel ZKAYA Fink Kurul Sekreteryasi

| Prof. Dr. Tayfun GÜLDÜR<br>Etik Kurul Başkanı | Rym Güldur. | | |
|---|---|---|---|
| Prof. Dr. Nigar VARDI<br>Etik Kurul Başkan Yrd. | KATILDI | Prof. Dr. Sermin TİMUR TAŞHAN<br>Etik Kurul Üyesi | KATILDI |
| Prof. Dr. Dinçer ÖZGÖR<br>Etik Kurul Üyesi | KATILDI | Prof. Dr. Serap PARLAR KILIÇ<br>Etik Kurul Üyesi | KATILDI |
| Prof. Dr. Ahmet KOÇ<br>Etik Kurul Üyesi | KATILDI | | |